CLINICAL TRIAL: NCT00002702
Title: Multicentre Randomised Trial of Inductive and Adjuvant Perilymphatically Injected Proleukin (rlL-2) in The Treatment of Operable Primary Squamous Cell Carcinoma of The Oral Cavity and Oropharynx
Brief Title: Surgery and Radiation Therapy With or Without Interleukin-2 in Treating Patients With Cancer of the Mouth or Oropharynx
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Institute of Oncology (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000064500; CNR-9506; EU-95024
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2011-02

CONDITIONS: Head and Neck Cancer
Keywords: stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — aldesleukin; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Biological: aldesleukin
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill cancer cells of the mouth or oropharynx. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not known whether giving interleukin-2 with surgery and radiation therapy is more effective than surgery and radiation therapy alone.

PURPOSE: This randomized phase III trial is studying surgery and radiation therapy alone to see how well they work compared to surgery, radiation therapy, and interleukin-2 in treating patients with cancer of the mouth or oropharynx.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free and overall survival in patients with previously untreated squamous cell carcinoma of the oral cavity or oropharynx treated with resection with or without and neoadjuvant and adjuvant perilymphatic interleukin-2 (IL-2) and radiotherapy.
* Compare the response rate in patients treated with these regimens.
* Determine the local and systemic effects of locoregional IL-2 on host-tumor interaction and immune properties in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center and tumor stage (T2, N0-2 vs T2, N3 or T3-4, N0-3). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo induction comprising interleukin-2 (IL-2) via perilymphatic injections to the ipsilateral myelohyoid muscle and insertion of the sternocleidomastoid muscle on days 1-5 and 8-12. Within 10 days after the last IL-2 injection, patients undergo en bloc resection of the primary tumor and corresponding lymphatic drainage area and pre-study margins. Beginning within 4 weeks after surgery, patients with T2, N0-3 disease but with pathohistological evidence of node invasion or capsular rupture of node metastasis or T3-4, N0-3 disease undergo adjuvant radiotherapy 5 days a week for 4.5-6.5 weeks. Beginning within 4 weeks after surgery or radiotherapy (if applicable), patients receive adjuvant IL-2 via perilymphatic injections to the contralateral myelohyoid muscle and insertion of the sternocleidomastoid muscle on days 1-5. Adjuvant IL-2 continues monthly for at least 1 year in the absence of disease progression.
* Arm II: Patients undergo resection and radiotherapy (if eligible) as in arm I. Patients are followed monthly for 1 year and then every 2 months for 2 years.

PROJECTED ACCRUAL: A total of 260 patients (130 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven squamous cell carcinoma of the oral cavity or oropharynx

  * Operable, primary, unilateral, stage T2-4, N0-3, M0 disease
  * No high probability of bilateral lymphatic spread (requirement for bilateral neck dissection)
* No tumor involvement of the following sites:

  * Pterygopalatine fossa
  * Carotid artery
  * Maxillary sinus
  * Facial skin
  * Anterior floor of the mouth
  * Base of the tongue infiltrating more than 1 cm
* Measurable or evaluable disease by physical exam and/or noninvasive imaging

PATIENT CHARACTERISTICS:

Age:

* 75 and under

Performance status:

* ECOG 0-2 OR
* Karnofsky 70-100%

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 4,000/mm3
* Platelet count at least 60,000/mm3
* Hematocrit at least 30%

Hepatic:

* Bilirubin normal
* Hepatitis B surface antigen negative

Renal:

* Creatinine normal

Cardiovascular:

* No congestive heart failure
* No uncontrolled hypertension
* No coronary artery disease
* No serious arrhythmia
* No evidence of prior myocardial infarction on ECG (stress test required if in doubt)

Other:

* HIV negative
* No autoimmune disease
* No contraindications to pressor agents
* No serious infection requiring antibiotics
* No other concurrent primary malignancy
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior or other concurrent immunotherapy

Chemotherapy:

* No prior or concurrent chemotherapy

Endocrine therapy:

* No prior or concurrent hormonal therapy
* No concurrent corticosteroids

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics
* No prior major organ allografts

Other:

* No other prior therapy
* No other concurrent investigational drugs, agents, or devices
* No concurrent nonsteroidal antiinflammatory drugs, ranitidine, cimetidine, or coumarin

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 1992-09

PRIMARY OUTCOMES:
Disease-free survival at 3 and 5 years
Recurrence/metastasis rate at 3 and 5 years
Response rate
Local and systemic effects of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Cortesina, MD, Study Chair — Universita Degli Studi di Turin
Locations (7):
- Italy (7):
  - Universita Degli Studi di Bari, Bari
  - Cattedra di Oncologia Medica - Universita degli Studi di Cagliari, Cagliari
  - Universita di Ferrara, Ferrara
  - Universita Degli Studi di Florence - Policlinico di Careggi, Florence
  - Universita di Torino, Turin
  - Azienda Sanitaria Ospedaliera Ordine Mauriziano, Turin
  - Ospedale San Bortolo, Vicenza